CLINICAL TRIAL: NCT03723070
Title: Cryterion Cardiac Cryoablation System CE Mark Study
Brief Title: Cryoablation System FIM/CE Mark Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Cryterion Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEM-A02-02
Record Dates: First submitted 2017-11-28; First posted 2018-10-29 (Actual); Results first posted 2021-07-19 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2021-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Non-randomized study designed to validate the safety and performance of the Cryterion Cardiac Cryoablation System when used as intended
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PV Cryoablation (Experimental): Ablation of the ostium of the pulmonary veins (PV) as a means to electrically isolate the veins in the treatment of atrial fibrillation. A cryoablation balloon will be inserted into the left atrium and cryo applications will be administered to create an endocardial thermal injury by using the Cryterion Cardiac Cryoablation System
  Interventions: Device: The Cryterion Cardiac Cryoablation System

INTERVENTIONS:
Device: The Cryterion Cardiac Cryoablation System — Cryoablation System that includes a Balloon Catheter, Circular Mapping Catheter, Steerable Sheath and Cryoablation Console. In combination, components of the System will be inserted into the left atrium and a thermal injury at the PV ostium will be created to electrically isolate the veins

SUMMARY:
Multi-center, open label, prospective clinical study to establish the acute safety and performance of the Cryterion Cardiac Cryoablation System

DETAILED DESCRIPTION:
This is a single-arm, open-label clinical study using a cryoablation balloon device to isolate pulmonary veins during an atrial fibrillation ablation procedure. Cryo is a scientifically proven energy source used to create a thermal injury during endocardial ablation. The investigational device uses current technology with minor design modifications and will be studied to validate similarities in the safety and performance parameters compared to literature.

ELIGIBILITY:
Main Inclusion Criteria:

* Currently scheduled for a de novo ablation of atrial fibrillation (AF) defined as AF with self-terminating episodes lasting no longer than 7 continuous days (PAF)

Main Exclusion Criteria:

* In the opinion of the Investigator, any known contraindication to an AF ablation, Transesophageal Echocardiogram (TEE). or anticoagulation
* Any duration of continuous AF lasting longer than 7 days
* History of previous left atrial ablation or surgical treatment for Atrial Fibrillation/Atrial Flutter/Atrial Tachycardia (AF/AFL/AT)
* More than four (4) electrical cardioversions in the year prior to enrollment excluding cardioversions performed within 24 hours of arrhythmia onset.
* Significant structural heart disease or implanted cardiac devices

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarfaraz Taher, Study Director — Boston Scientific Corporation
Locations (4):
- Clinical Hospital Centre Split, Split, Croatia
- Netherlands (2):
  - Catharina Ziekenhuis, Eindhoven
  - Erasmus MC, Rotterdam
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anic A, Lever N, Martin A, Breskovic T, Sulkin MS, Duffy E, Saliba WI, Niebauer MJ, Wazni OM, Varma N. Acute safety, efficacy, and advantages of a novel cryoballoon ablation system for pulmonary vein isolation in patients with paroxysmal atrial fibrillation: initial clinical experience. Europace. 2021 Aug 6;23(8):1237-1243. doi: 10.1093/europace/euab018. PMID 33729470
- [Result] Martin A, Fowler M, Breskovic T, Ouss A, Dekker L, Yap SC, Bhagwandien R, Albrecht EM, Cielen N, Richards E, Tran BC, Lever N, Anic A. Novel cryoballoon to isolate pulmonary veins in patients with paroxysmal atrial fibrillation: long-term outcomes in a multicentre clinical study. J Interv Card Electrophysiol. 2022 Dec;65(3):609-616. doi: 10.1007/s10840-022-01200-5. Epub 2022 Apr 12. PMID 35412168

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PV Cryoablation
Started | 88
Completed | 79
Not Completed | 9
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 1
Not completed — Ended the study at 1 month follow-up visit as per applicable protocol at that time | 6

BASELINE CHARACTERISTICS:
Arm/Group | PV Cryoablation
Number analyzed (Participants) | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 81
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  New Zealand | 15
  Netherlands | 9
  Croatia | 64

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Outcome: Percentage of Participants With Procedure Related Adverse Events OR Device Related Adverse Events OR Serious Adverse Device Effects
Description: Percentage of participants with procedure related adverse events OR device related adverse events OR Serious Adverse device effects including: Death, Myocardial Infarction, Cardiac perforation/pericardial tamponade, Cerebral Infarct or systemic embolism, Major bleeding requiring transfusion of blood products, Mitral or tricuspid valvular damage, phrenic nerve damage causing persistent diaphragmatic paralysis, Symptomatic pulmonary vein stenosis, atrio-esophageal fistula, Air embolism leading to life-threatening event, other serious adverse device effects (SADEs)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | PV Cryoablation
Number analyzed (Participants) | 88
Participants | 50

2. Primary Outcome: Acute Procedural Success
Description: Percentage of patients achieving pulmonary vein isolation defined as entrance and exit block for each of the targeted pulmonary veins following the last ablation application.
Time Frame: Following the last cryo-application for each of the targeted veins, during the index procedure. Mean procedure time was 118 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | PV Cryoablation
Number analyzed (Participants) | 88
Participants | 87

3. Primary Outcome: 12 Month Treatment Success - Percentage of Subjects Free From Arrhythmias at 12 Months
Description: A treatment failure is defined as a subject being an acute procedural failure, having more than one repeat procedure during the 90-day blanking period or having a documented, symptomatic episode(s) of atrial fibrillation or atrial tachycardia, between 91 and 365 days post index procedure. Occurrence or recurrence of a right atrial arrhythmia is not considered a treatment failure post the 90-day blanking period
Time Frame: 12 months
Population: In total, 88 subjects were enrolled. Six subjects ended the study at the one month follow-up visit and were therefore not eligible for the analysis. Of the 3 subjects that were withdrawn prior to study completion, one subject experienced a recurrence before being withdrawn and was therefore included in the analysis. The two other subjects were event free at time of study withdrawal.
Measure: Count of Participants; unit: Participants
Arm/Group | PV Cryoablation
Number analyzed (Participants) | 80
Participants | 58

4. Secondary Outcome: Secondary Safety Outcome: Number of Procedure-related or Device Related Adverse Events.
Description: All procedure-related or device related adverse events with causal relationship
Time Frame: 12 months
Population: Causally related to procedure
Measure: Number; unit: Adverse Events
Arm/Group | PV Cryoablation
Number analyzed (Participants) | 88
Adverse Events | 12

5. Secondary Outcome: Percentage of Subjects With Isolation Immediately Post Ablation and With Reconnection During the Entrance/Exit Block Testing
Description: Percentage of subjects that present PV isolation immediately after ablation but show reconnection after 30 minutes during entrance/exit block testing.
  This outcome is only measured in subjects that were enrolled under the protocol that required a 30 minute waiting period between isolation and verification of isolation.
Time Frame: 30 minutes
Population: Out of 88 subjects enrolled in the study, 54 subjects have been enrolled under the protocol requiring a 30 minute waiting period between pulmonary vein isolation and entrance/exit block testing. All subjects for whom at least one additional application was performed minimally 30 minutes after the previous ablation, were considered having a potential reconnection during entrance/exit block testing.
Measure: Count of Participants; unit: Participants
Arm/Group | PV Cryoablation
Number analyzed (Participants) | 54
Participants | 7

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | PV Cryoablation
All-Cause Mortality (participants affected / at risk) | 0/88
Serious Adverse Events (participants affected / at risk) | 6/88
Other Adverse Events (participants affected / at risk) | 56/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PV Cryoablation (N=88)
Episodic aphasia (Nervous system disorders) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 1 (1)
Cholelithiasis (Gastrointestinal disorders) | 1 (1)
Embolism in right femoral artery (Vascular disorders) | 1 (1)
Atrial Arrhythmia (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PV Cryoablation (N=88)
Post surgical wound discomfort (Skin and subcutaneous tissue disorders) | 2 (2)
Minor oozing/bleeding (Vascular disorders) | 3 (3)
Angina/Chest pain (Cardiac disorders) | 4 (5)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Hematoma (Skin and subcutaneous tissue disorders) | 3 (3)
Nerve (weakness, palsy) (Nervous system disorders) | 4 (4)
Adverse reactions (General disorders) | 1 (1) — Intermittent fever and coughing
Adverse reaction - hypotension (Cardiac disorders) | 3 (3)
Adverse reaction - neurological (Nervous system disorders) | 1 (1) — Migraine
Adverse reaction Anesthesia/sedation (Gastrointestinal disorders) | 2 (2) — Nausea
Adverse reaction - gastrointestinal (Gastrointestinal disorders) | 3 (3) — Gastric reflux, vomitting, nausea
Adverse reaction - pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Dyspnea
Sore Throat post procedure (Injury, poisoning and procedural complications) | 1 (1)
Palpitations (Cardiac disorders) | 27 (38)
Atrial Arrhythmia (Cardiac disorders) | 10 (11)
Syncope (Cardiac disorders) | 1 (1)
Diziness (Cardiac disorders) | 2 (2)
Chest Pain (Cardiac disorders) | 3 (3)
Dyspnea (Cardiac disorders) | 1 (1)
Fatigue/Weakness (Cardiac disorders) | 3 (3)
Inability to palpate peripheral arterial pulse (Cardiac disorders) | 1 (1)
CVA (Cardiac disorders) | 1 (1)
Adverse Reaction - Urticaria (General disorders) | 1 (1)
Adverse Reaction - Medication (General disorders) | 1 (1)
Hipoechogenic lesion in left breast (General disorders) | 1 (1)
Fever - Virus (Infections and infestations) | 3 (3)
Ankle Injury (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypersaturation with warfarin (Blood and lymphatic system disorders) | 1 (1)
Elevated level Thyroid function (T4) (Endocrine disorders) | 1 (1)
Infection (Infections and infestations) | 1 (2)
Shinlges (Nervous system disorders) | 1 (1) — Rash due to shingles (viral infection that causes a painful rash) on the back
Gastritis (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Polipectomy (Gastrointestinal disorders) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Polyp in acsending colon (Gastrointestinal disorders) | 1 (1)
Urinary Infection (Renal and urinary disorders) | 1 (1)
Positive urine culture (Renal and urinary disorders) | 1 (1)
Benign renal cyst L) kidney (Renal and urinary disorders) | 1 (1)
Muskuloskeletal (Musculoskeletal and connective tissue disorders) | 3 (3) — Chest and neck pain, knee pain,
Pharyngitis (Infections and infestations) | 1 (1)
Epistaxis (Vascular disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Conjunctavitis (Eye disorders) | 1 (1)
Type 2 Diabetes Mellitus (Endocrine disorders) | 1 (1)
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haematoma of the right upper arm (Skin and subcutaneous tissue disorders) | 1 (1)
sinusitis (Infections and infestations) | 1 (1)
Tooth Pain (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/70/NCT03723070/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT03723070/SAP_001.pdf